CLINICAL TRIAL: NCT02111278
Title: Lumbar Manipulation and Exercise for the Treatment of Acute Low Back Pain in Adolescents: a Randomized Controlled Trial
Brief Title: Lumbar Manipulation and Exercise for the Treatment of Acute Low Back Pain in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Research Coordinator, Sports and Orthopedic Physical Therapy Department, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB11-00262
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Low Back Pain
Keywords: Manipulation; Lumbar; Low Back Pain; Manual Therapy; Adolescents
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lumbar Manipulation (Experimental): Patients randomized to this treatment group will receive lumbar manipulation during the first 2 physical therapy visits. Patient will receive 4 weeks of physical therapy 2 visits per week.
  Interventions: Other: Lumbar Manipulation; Other: Physical Therapy
- Sham Manipulation (Placebo Comparator): Patients randomized to this treatment group will receive a sham manipulation during the first 2 physical therapy visits. Patient will receive 4 weeks of physical therapy 2 visits per week.
  Interventions: Other: Sham Manipulation; Other: Physical Therapy

INTERVENTIONS:
Other: Lumbar Manipulation — The manipulating therapist performs the lumbar manipulation technique. With the patient supine, the therapist stands opposite the side to be manipulated. The patient is passively side-bent away from the therapist. The therapist rotates the thoracic spine and then delivers a quick posterior and inferior thrust through the anterior superior iliac spine. The manipulation is performed on the side the patient reported to be more symptomatic. If the patient is unable to identify a more painful side, the side to be manipulated is left to the manipulating therapist discretion. If a cavitation is experienced, no more manipulations are performed that session. If no cavitation is produced, the patient is repositioned, and the manipulation is attempted again. If no cavitation is experienced again, the therapist attempts to manipulate the opposite side. A maximum of two attempts per side will be attempted.
  Arms: lumbar Manipulation
Other: Sham Manipulation — The manipulating therapist will perform the sham lumbar manipulation technique with the patient side-lying. The therapist passively flexes both hips until slight lumbar flexion is noted at the patient's most painful vertebral level. The therapist will take time palpating patient's spine taking care to avoid rotating the spine. The therapist will then place both hands on the same lumbar spinous process. An equal and opposite force is then applied to the spinous process with both hands. No physiologic motion is expected with this technique. The patient will then be setup for the same sham technique on the opposite side. The sham manipulation technique will be performed in an attempt to blind the patient to group allocation. This technique is designed to provide similar hands on treatment time as the manipulation intervention.
  Arms: Sham Manipulation
Other: Physical Therapy — Patients will receive 4 weeks of physical therapy with 2 visits per week. The treating physical therapist is blinded to group allocation. The treating physical therapist will prescribe exercises based on patient presentation. Therapy visits last approximately 45-60 minutes depending of patient ability to perform exercises. The treating physical therapist will perform no mobilizations or manipulations on the patient.

SUMMARY:
The purpose of this study is to determine if the addition of lumbar manipulation will improve function, decrease pain, and recurrence in adolescents with low back pain. The secondary aim of this study is to determine if a modification of a clinical prediction rule by Flynn will be effective in identifying adolescent patients with low back pain who would benefit from lumbar manipulation.

DETAILED DESCRIPTION:
This is a double blind, randomized controlled, parallel group study. The investigators will consider adolescent patients with a primary complaint of low back pain referred to physical therapy.

The purpose of this study is to determine if the addition of lumbar manipulation will improve function, decrease pain, and recurrence in adolescents with low back pain. The secondary aim of this study is to determine if a modification of a clinical prediction rule by Flynn will be effective in identifying adolescent patients with low back pain who would benefit from lumbar manipulation.

Prior to randomization, patients will complete several self-report measures and then receive a standardized history and physical examination performed by the treating physical therapist. The information collected will include age, sex, duration and nature of symptoms. Standardized physical examination measures include lumbar active range of motion assessment for quality and mobility, lumbar segmental mobility, hip internal rotation range of motion, straight leg raise test, and prone instability test. Treating physical therapists were trained in all evaluation measures before data collection began. Patients are assessed on each item of a modified clinical prediction rule which consists of 4 items; duration of symptoms, symptoms distal to knee, Hip Internal Rotation >35 degrees, and presence of lumbar segmental hypomobility. The fear avoidance beliefs questionnaire work sub-scale component was removed since the score would likely not be valid in the adolescent population. Meeting 3 of the 4 items was considered to be positive on the rule in this population.

The manipulating therapist who performs the intervention will be aware of treatment allocation, whereas the treating physical therapist and patients are blinded to treatment group allocation. To assess if the patients are successfully blinded to group allocation, the investigator will ask each patient to guess which intervention was performed on them following discharge from therapy.

Randomization is determined by checking a randomly generated computer list that tells the manipulating therapist the assigned group. The computer list was generated by an aide not involved in the study who blindly drew 52 cards that placed an equal number of patients into either the manipulation or sham group.

To address the issue of safety, patients who experience a clinically significant decrease in functional ability or increase in pain will be classified as having an adverse reaction. The minimally clinical important difference for the Patient Specific Functional Scale is >= 6. While the minimal clinical important difference of the Numeric Pain Rating Scale is 2 points. Following the manipulation or sham intervention patients will be asked if they experienced pain or discomfort during or following the intervention. An interim analysis is planned at the midpoint of the study to assess the safety and efficacy of the intervention. If >1/3 of patients in the manipulation group have a worsening of symptoms at any follow up, the study will be terminated for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* patients 13 to 17 years old
* duration of low back symptoms less than 90 days

Exclusion Criteria:

* contraindication to manipulation. These included "red flags" for physical therapy, previous lumbar surgery, those who had signs consistent with nerve root compression (positive straight-leg test of < 45 degrees, diminished reflexes, sensation, or lower extremity strength), those who were pregnant, and those diagnosed with, or suspected of having a spondylolysis or spondylolisthesis.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Patient Specific Functional Scale | Initial Evaluation, 1 week, 4 weeks, and 6 month
  The Patient Specific Functional scale asks the participant to nominate 3 important activities they are not able to do or are having difficulty performing because of their back pain. Each activity is scored on a numerical rating scale from 0 (unable to perform) to 10 (able to perform at pre-injury level).

SECONDARY OUTCOMES:
Global Rating of Change scale | 1 week, and 4 weeks
  The Global Rating of Change scale is a 15-point Likert type scale (-7 to +7). A score of 0 represents no change from initial injury, +7 represents a great deal better, and -7 represents a great deal worse.
Change in Numeric Pain Rating Scale | Initial Evaluation, 1 week, 4 weeks, and 6 month
  The Numeric Pain Rating Scale is an 11-point pain-rating scale ranging from 0 (no pain) to 10 (worst imaginable pain) to assess current pain intensity and the best and worst level of pain during the last 24 hours. An average of the 3 ratings will be used.

OTHER OUTCOMES:
Recurrence of low back pain | 6 months
  Patients will be asked if they have had significant pain or a recurrence of pain in the low back since therapy has ended. Yes or No response from the patient.
Sought further treatment | 6 months
  Patient will be asked if they sought further treatment for their low back pain after 4 weeks of physical therapy ended.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C Selhorst, DPT, Principal Investigator — Nationwide Children's Hospital
Locations (3):
- United States (3):
  - Nationwide Children's Hospital Sports and Ortho PT Ortho Center, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Westerville, Westerville, Ohio

REFERENCES:
- [Background] Vaughn DW, Kenyon LK, Sobeck CM, Smith RE. Spinal manual therapy interventions for pediatric patients: a systematic review. J Man Manip Ther. 2012 Aug;20(3):153-9. doi: 10.1179/2042618612Y.0000000007. PMID 23904755
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Ndetan H, Evans MW Jr, Hawk C, Walker C. Chiropractic or osteopathic manipulation for children in the United States: an analysis of data from the 2007 National Health Interview Survey. J Altern Complement Med. 2012 Apr;18(4):347-53. doi: 10.1089/acm.2011.0268. Epub 2012 Mar 2. PMID 22384933
- [Background] Koppenhaver SL, Fritz JM, Hebert JJ, Kawchuk GN, Childs JD, Parent EC, Gill NW, Teyhen DS. Association between changes in abdominal and lumbar multifidus muscle thickness and clinical improvement after spinal manipulation. J Orthop Sports Phys Ther. 2011 Jun;41(6):389-99. doi: 10.2519/jospt.2011.3632. Epub 2011 Apr 6. PMID 21471653
- [Background] Vela LI, Haladay DE, Denegar C. Clinical assessment of low-back-pain treatment outcomes in athletes. J Sport Rehabil. 2011 Feb;20(1):74-88. doi: 10.1123/jsr.20.1.74. PMID 21411824
- [Background] Wang YC, Hart DL, Stratford PW, Mioduski JE. Baseline dependency of minimal clinically important improvement. Phys Ther. 2011 May;91(5):675-88. doi: 10.2522/ptj.20100229. Epub 2011 Mar 3. PMID 21372203
- [Background] Fritz JM, Koppenhaver SL, Kawchuk GN, Teyhen DS, Hebert JJ, Childs JD. Preliminary investigation of the mechanisms underlying the effects of manipulation: exploration of a multivariate model including spinal stiffness, multifidus recruitment, and clinical findings. Spine (Phila Pa 1976). 2011 Oct 1;36(21):1772-81. doi: 10.1097/BRS.0b013e318216337d. PMID 21358568
- [Background] Stanton TR, Fritz JM, Hancock MJ, Latimer J, Maher CG, Wand BM, Parent EC. Evaluation of a treatment-based classification algorithm for low back pain: a cross-sectional study. Phys Ther. 2011 Apr;91(4):496-509. doi: 10.2522/ptj.20100272. Epub 2011 Feb 17. PMID 21330450
- [Background] Hall AM, Maher CG, Latimer J, Ferreira ML, Costa LO. The patient-specific functional scale is more responsive than the Roland Morris disability questionnaire when activity limitation is low. Eur Spine J. 2011 Jan;20(1):79-86. doi: 10.1007/s00586-010-1521-8. Epub 2010 Jul 14. PMID 20628767
- [Background] Humphreys BK. Possible adverse events in children treated by manual therapy: a review. Chiropr Osteopat. 2010 Jun 2;18:12. doi: 10.1186/1746-1340-18-12. PMID 20525194
- [Background] Fritz JM, Clifford SN. Low back pain in adolescents: a comparison of clinical outcomes in sports participants and nonparticipants. J Athl Train. 2010 Jan-Feb;45(1):61-6. doi: 10.4085/1062-6050-45.1.61. PMID 20064050
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Resnik L, Liu D, Mor V, Hart DL. Predictors of physical therapy clinic performance in the treatment of patients with low back pain syndromes. Phys Ther. 2008 Sep;88(9):989-1004. doi: 10.2522/ptj.20070110. Epub 2008 Aug 8. PMID 18689610
- [Background] Chen KC, Chiu EH. Adolescent idiopathic scoliosis treated by spinal manipulation: a case study. J Altern Complement Med. 2008 Jul;14(6):749-51. doi: 10.1089/acm.2008.0054. PMID 18673077
- [Background] Vohra S, Johnston BC, Cramer K, Humphreys K. Adverse events associated with pediatric spinal manipulation: a systematic review. Pediatrics. 2007 Jan;119(1):e275-83. doi: 10.1542/peds.2006-1392. Epub 2006 Dec 18. PMID 17178922
- [Background] Childs JD, Flynn TW, Fritz JM. A perspective for considering the risks and benefits of spinal manipulation in patients with low back pain. Man Ther. 2006 Nov;11(4):316-20. doi: 10.1016/j.math.2005.09.002. Epub 2006 Jul 12. PMID 16839800
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Childs JD, Fritz JM, Flynn TW, Irrgang JJ, Johnson KK, Majkowski GR, Delitto A. A clinical prediction rule to identify patients with low back pain most likely to benefit from spinal manipulation: a validation study. Ann Intern Med. 2004 Dec 21;141(12):920-8. doi: 10.7326/0003-4819-141-12-200412210-00008. PMID 15611489
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] O'Neal ML. The pediatric spine: anatomical and dynamic considerations preceding manipulation. Compr Ther. 2003 Summer-Fall;29(2-3):124-9. doi: 10.1007/s12019-003-0016-5. PMID 14606342
- [Background] Clifford SN, Fritz JM. Children and adolescents with low back pain: a descriptive study of physical examination and outcome measurement. J Orthop Sports Phys Ther. 2003 Sep;33(9):513-22. doi: 10.2519/jospt.2003.33.9.513. PMID 14524510
- [Background] McNeely ML, Torrance G, Magee DJ. A systematic review of physiotherapy for spondylolysis and spondylolisthesis. Man Ther. 2003 May;8(2):80-91. doi: 10.1016/s1356-689x(02)00066-8. PMID 12890435
- [Background] Flynn T, Fritz J, Whitman J, Wainner R, Magel J, Rendeiro D, Butler B, Garber M, Allison S. A clinical prediction rule for classifying patients with low back pain who demonstrate short-term improvement with spinal manipulation. Spine (Phila Pa 1976). 2002 Dec 15;27(24):2835-43. doi: 10.1097/00007632-200212150-00021. PMID 12486357
- [Background] Burton AK, Clarke RD, McClune TD, Tillotson KM. The natural history of low back pain in adolescents. Spine (Phila Pa 1976). 1996 Oct 15;21(20):2323-8. doi: 10.1097/00007632-199610150-00004. PMID 8915066